CLINICAL TRIAL: NCT05508360
Title: "Lumbar Operatively Inserted PerQdisc Artificial Implant Following Nulcectomy" (LOPAIN2)
Acronym: LOPAIN2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spinal Stabilization Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LOPAIN2
Record Dates: First submitted 2022-08-01; First posted 2022-08-19 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Degenerative Disc Disease; Chronic Low-back Pain
Keywords: Degenerative Disc Disease; DDD; Chronic Low Back Pain; cLBP; Disc Herniation; Nucleus Replacement; Low Back Pain
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral Disc Displacement; Low Back Pain

STUDY DESIGN:
Intervention Model Description: This is an open-label study. Patients will receive one implant if they meet all inclusion/exclusion criteria after a review by the Medical Advisory Board (MAB).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lumbar Disc Nucleus Replacement (Experimental): All patients meeting all inclusion criteria and no exclusion criteria will be considered for nucleus replacement surgery following a review by the Medical Advisory Board.
  Interventions: Device: PerQdisc Nucleus Replacement System

INTERVENTIONS:
Device: PerQdisc Nucleus Replacement System — Lumbar spine disc nucleus replacement system. All patients meeting all inclusion criteria and no exclusion criteria will be considered for nucleus replacement surgery following a review by the Medical Advisory Board.

SUMMARY:
This study will be a prospective, open-label, multi-center study including 72 patients that will collect additional safety and efficacy data for the Spinal Stabilization Technologies PerQdisc Nucleus Replacement System.

DETAILED DESCRIPTION:
This study will be a prospective, open-label, multi-center study that will collect additional safety and efficacy data for the minimally invasive PerQdisc Nucleus Replacement Device (NRD). Patients will have degenerative disc disease (DDD) in one or more lumbar discs. The NRD is used for surgical replacement of a single nucleus pulposus between spinal lumbar discs L1-S1 using any standard anterior, standard lateral, or minimally invasive posterolateral surgical approach. Currently the surgical gold standard involves spinal fusion of the affected vertebral bodies, reducing range of motion and increasing stress on other vertebral bodies. The goal of nucleus replacement is to reduce chronic low back pain by maintaining disc height while preserving range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Patient is skeletally mature aged 22-70.
* Patient has Degenerative Disc Disease (DDD) at one or more levels between L1 and S1 but the discogenic pain must be limited to a single level.
* Patient has adequate disc height (6mm) at the level to be treated
* Patient has exhausted a minimum of 6 months of conservative treatment for their back (e.g. physical therapy, medications, injections, life style changes, etc).
* Patient has a preoperative Oswestry Disability questionnaire score ≥ 40 out of 100 points (40/100)
* Patient has a low back pain Visual Analog Scale (VAS) ≥ 40 mm (4 cm)
* Patient has signed the approved Informed Consent Form.
* All surgeries must be approved by the Medical Advisory Board (MAB)

Exclusion Criteria:

* Patient has less than 6 mm of disc height.
* Patient has had prior lumbar spine surgery (nucleoplasty at non-index level is considered acceptable).
* Patient has had spinal fusion in the lumbar or thoracic intervertebral spaces. Cervical fusion is allowed as long as there are no neurologic deficits in the lower extremities.
* Patient has spondyloarthropathy or other spondylolisthesis greater than 2 mm.
* Patient has congenital moderate or severe spinal stenosis or epidural lipomatosis.
* Patient has significant facet disease. Significant is defined as pain improvement of 80% or more following image-guided medial branch blocks of the target level according to SIS guidelines (diagnostic, contrast controlled).
* Patient has any known active malignancy.
* Patient has previously undergone or currently on immunosuppressive therapy. Steroids used to treat inflammation are allowed.
* Patient has active or local systemic infection.
* Patient has been diagnosed with hepatitis, rheumatoid arthritis, lupus erythematosus, or other autoimmune disease including AIDS, ARC and HIV.
* Patient has diabetes mellitus (Type 1 or 2) requiring daily insulin management.
* Patient has osteopenia of the spine (T-score of -1.0 or lower). A DEXA scan should be performed to rule out patients considered at risk for osteopenia.
* Patient has morbid obesity defined as a body mass index (BMI) more than 40 or a weight of more than 45 kg (100 lbs.) over ideal body weight.
* Patient has a known allergy to silicone or barium sulfate.
* Patient has a significant disc herniation at the level to be treated. Significant is defined as a large, extruded herniation that creates a risk for expulsion.
* Patient has a significant Schmorl's node in the level to be treated. Significant is defined as a large, rectangular or irregular shaped node that has an associated active inflammatory process (Modic I changes).
* Patient has motion of less than 3 degrees on pre-operative lateral flexion/extension radiographs.
* Patient belongs to a vulnerable population or has a condition such that his/her ability to provide informed consent, comply with follow-up requirements, or provide self-assessments is compromised (e.g. developmentally, disabled, prisoner, chronic alcohol/ substance abuser)

Intraoperative Exclusion Criteria:

* Protrusion of the 20A Imaging Balloon up to or beyond the outer margin of the vertebra during the imaging steps.
* Patient has a violated endplate as determined by imaging balloons during fluoroscopy.
* Patient has a disc space that is too narrow for implantation. MIPL Specific
* Poor radiological visualization of Kambin's triangle.
* Sustained irritation of the exiting nerve root during any aspect of the annular dilation technique (leg movement or if performing with electrical monitoring) in spite or repositioning instruments.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2027-08-22 (Estimated); Study Completion 2030-08-22 (Estimated)

PRIMARY OUTCOMES:
Perfromance: ODI | 6 months
  Change in in Oswestry Disability Index (ODI) comparing baseline to follow up visits using a patient-reported outcome tool
Perfromance: ODI | 12 months
  Change in in Oswestry Disability Index (ODI) comparing baseline to follow up visits using a patient-reported outcome tool
Performance: VAS | 6 months
  Change in back pain as measured by the 100 - millimeter Visual Analog Scale (VAS)
Performance: VAS | 12 months
  Change in back pain as measured by the 100 - millimeter Visual Analog Scale (VAS)
Safety: Expulsion & Device Failure | 6 months
  Incidence of device expulsion and device failure following surgery based on follow up X-rays and MRI's
Safety: Expulsion & Device Failure | 12 months
  Incidence of device expulsion and device failure following surgery based on follow up X-rays and MRI's

SECONDARY OUTCOMES:
Safety: Revision Surgery | 6 months, 12 months, and 5 years
  Incidence of revision surgery
Safety: Expulsion & Device Failure | 5 years
  Incidence of device expulsion and device failure following surgery based on follow up X-rays and MRI's
Performance: Disc Height | 6 months, 12 months, and 5 years
  Preservation of intervertebral disc height (in mm) as measured on MRI post-surgery compared to baseline
Performance: RoM | 6 months, 12 months, 5 years
  Preservation of range of movement (expressed in degrees) at the index and adjacent levels at baseline compared to follow-up using flexion/extension radiographs
Safety: Neurological Status | 6 months, 12 months, and 5 years
  Maintenance of baseline neurologic status through physical assessment evaluating nerve compression at baseline and post-surgical follow-up using pain, motor strength, and sensation feedback from the patient on a 0 (no compression) to 5 (major compression) scale
Performance: Analgesic Score | 6 months, 12 months, and 5 years
  Change in level of pain medication used comparing baseline to follow up visits based on a medication scale ranging from 0 (no meds) - 4 (high dose opioids)
Safety: SAE | 6 months, 12 months, and 5 years
  Incidence of serious adverse events that are related to the surgical procedure or Incidence of Serious Adverse Events related to the surgical procedure or device

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Golan, MD, Study Chair — Jewish General Hospital; Michael Hess, MD, Study Chair — London Spine Clinic/ATOS-Klinik
Locations (10):
- Colombia (7):
  - CIGE: Centro de Imunologia y Genetica, Medellín, Antioquia
  - Fundacion Hospitalaria San Vicente de Paul, Medellín, Antioquia
  - Cediul S.A., Barranquilla, Atlántico
  - Fundación Campbell, Barranquilla, Atlántico
  - Sabbag Radiólogos S.A., Barranquilla, Atlántico
  - Sociedad de Cirugia de Bogota- Hospital de San Jose, Bogotá, D.C.
  - Clínica Imbanaco de Cali S.A., Cali, Valle del Cauca Department
- Pacífica Salud Hospital Punta Pacífica, Panama City, Provincia de Panamá, Panama
- Sanatario Americano, Asunción, Paraguay
- Republican Specialized Scientific Practical Medical Center of Endocrinology named after Academician Y.Kh. Turakulova, Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: No